CLINICAL TRIAL: NCT02480114
Title: A Randomized Phase III Trial of Gabapentin Versus Standard of Care for Prevention and Treatment of Mucositis in Locally Advanced Head and Neck Cancer Patients Undergoing Primary or Adjuvant Chemoradiation
Brief Title: Gabapentin Compared to Standard of Care in Preventing Mucositis in Patients With Stage III-IV Head and Neck Cancer Undergoing Primary or Adjuvant Chemoradiation Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Derek Smith, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC HN 1541; NCI-2015-00750 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VICC HN 1541 (Other: Vanderbilt University/Ingram Cancer Center); P30CA068485 (NIH)
Record Dates: First submitted 2015-06-16; First posted 2015-06-24 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-01

CONDITIONS: Malignant Head and Neck Neoplasm; Mucositis; Radiation-Induced Disorder
MeSH Terms: conditions — Head and Neck Neoplasms; Mucositis; Abnormalities, Radiation-Induced | interventions — Early Intervention, Educational; Educational Status; Methods; Gabapentin; cyclohexaneacetic acid; Analgesia; Pain Management; oxycodone-acetaminophen; acetaminophen, hydrocodone drug combination; Fentanyl; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I Standard of Care (Active Comparator): Patients receive standard of care consisting of oral health measures, oral rinsing, miracle mouthwash, nonsteroidal anti-inflammatories, and opioid analgesics. Patients also undergo an education session at the beginning of treatment to review foundations of oral care and pain management.
  Interventions: Other: Educational Intervention; Other: Pain Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Oxycodone/Acetaminophen; Drug: Hydrocodone/Acetaminophen; Drug: Fentanyl; Drug: Ibuprofen; Drug: Magic Mouthwash
- Arm II Standard of Care Plus Gabapentin (Experimental): Patients receive standard of care and undergo an education session as in Arm I. Patients also receive gabapentin PO three times a day throughout chemoradiation treatment (approximately 5-7 weeks) and until mucositis resolves and pain subsides.
  Interventions: Other: Educational Intervention; Drug: Gabapentin; Other: Pain Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Oxycodone/Acetaminophen; Drug: Hydrocodone/Acetaminophen; Drug: Fentanyl; Drug: Ibuprofen; Drug: Magic Mouthwash

INTERVENTIONS:
Other: Educational Intervention — Undergo oral care and pain management education session
  Other Names: Education for Intervention
Drug: Gabapentin — Given PO
  Other Names: Gralise; Neurontin; 1-(aminomethyl) cyclohexaneacetic Acid, 60142-96-3,
  Arms: Arm II Standard of Care Plus Gabapentin
Other: Pain Therapy — Receive usual oral health care
  Other Names: Analgesia; Pain Control; Pain Management; Pain
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Oxycodone/Acetaminophen — Analgesia
  Other Names: Percocet
Drug: Hydrocodone/Acetaminophen — Analgesia
  Other Names: Lortab; Vicodin
Drug: Fentanyl — Transdermal Analgesia
  Other Names: Duragesic
Drug: Ibuprofen — NSAID Analgesia
  Other Names: Motrin; Advil
Drug: Magic Mouthwash — Oral Solution to treat mucositis
  Other Names: Miracle Mouthwash; First-Mouthwash BLM; First-BXN Mouthwash

SUMMARY:
This randomized phase III trial studies how well gabapentin plus standard of care work compares to standard of care without Gabapentin in preventing inflammation of the mucous membranes (mucositis) in patients with stage III-IV head and neck cancer that are undergoing primary or subsequent (adjuvant) chemoradiation therapy. Radiation therapy to the head and neck may cause a burn involving the inside of the mouth, throat, and nasal passages, resulting in pain. Gabapentin may help prevent (or minimize) pain associated with radiation-induced mucositis in patients with head and neck cancer.

DETAILED DESCRIPTION:
Primary Objectives:

- To determine whether gabapentin used as a preventive measure during chemoradiation can reduce radiation-induced mucositis associated pain in head and neck cancer patients as measured by: 1) pain scores on the Vanderbilt Head and Neck Symptom Survey (VHNSS version 2.), and 2) analgesic use.

Secondary Objectives:

* To assess the safety (grade 3 or 4 adverse events) and tolerability of using gabapentin (discontinuation of drug due to side effects - yes or no)
* To correlate pain severity with frequency and severity of general systemic symptoms.

Exploratory Objectives:

- To determine whether pain control is associated with weight loss (in pounds) and duration of use of percutaneous endoscopic gastrostomy utilization (in days).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Standard of Care (usual care) - Patients receive consisting of oral health measures, oral rinsing, miracle mouthwash, nonsteroidal anti-inflammatories, and opioid analgesics. Patients also undergo an education session at the beginning of chemoradiation treatment to review foundations of oral care and pain management.

ARM II: Standard of Care plus Gabapentin - Patients receive standard of care and undergo an education session as in Arm I. Patients also receive gabapentin orally (PO) three times a day throughout chemoradiation treatment (approximately 5-7 weeks) and until mucositis resolves and pain subsides.

After completion of study treatment, patients are followed up monthly for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven cancer of the head and neck cancer
* Stage 3 or 4
* Planned primary or adjuvant chemoradiation therapy
* Willing and able to provide informed consent
* English speaking

Exclusion Criteria:

* Currently on gabapentin
* Prior non-tolerance of gabapentin
* History of seizure disorder

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-07; Primary Completion 2019-09 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Smith, DDS,PhD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Vanderbilt Medical Center in Nashville, TN from July 2015 to May 2019. 79 participants were recruited and 8 of those withdrew.
Period: Overall Study
Arm/Group | Arm II Standard of Care Plus Gabapentin | Arm I Standard of Care
Started | 41 | 38
Completed | 32 | 30
Not Completed | 9 | 8
Not completed — Not completing surveys | 3 | 2
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Disease progression | 3 | 0
Not completed — Improper completion of survey | 1 | 1
Not completed — Not eligible | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I Standard of Care | Arm II Standard of Care Plus Gabapentin | Total
Number analyzed (Participants) | 38 | 41 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 34 | 66
  >=65 years | 6 | 7 | 13
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 61.5 [54.75 to 66.25] | 61 [52 to 66] | 61 [53 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 26 | 27 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 33 | 39 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 38 | 41 | 79

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Associated With Radiation-induced Mucositis, (Pain Subscale of the Vanderbilt Head and Neck Symptom Survey (VHNSS))
Description: The pain subscale is composed of 4 items of the Vanderbilt Head and Neck Symptom Survey. The subscale score was calculated by taking the first non-negative principle component of the 4 items. The scale was scores range from 0 to 10 with 10 representing the worst pain.
Time Frame: Up to 3 months post-treatment
Population: Longitudinal analysis was completed including all patients in both arms of the study. Although some patients stopped filling out surveys part way through the study and therefore are not marked as 'complete' in the patient flow section, the data they did provide was still used for analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm I Standard of Care | Arm II Standard of Care Plus Gabapentin
Number analyzed (Participants) | 32 | 39
score on a scale | 4.26 [3.98 to 5.16] | 3.68 [2.04 to 3.68]
Statistical Analysis 1: Comparison: Arm I Standard of Care vs Arm II Standard of Care Plus Gabapentin; Test type: Superiority; p = 0.004, Proportional Odds Regression; Odds Ratio (OR) = 0.549, 95% CI 2-sided [0.364 to 0.827]

2. Secondary Outcome: Number of Participants With Grade 3 or 4 Adverse Events, (Graded Using Common Terminology Criteria for Adverse Events Criteria 4.0)
Description: Graphical and descriptive statistical summaries will be generated. Mixed-level general linear modeling will be used. All tests of statistical significance will maintain maximum Type I error of 0.05 (p < 0.05). Frequency distributions will summarize the safety outcome.
Time Frame: Up to 3 months post-treatment
Population: All patients in both arms were analyzed. Although some patients stopped filling out surveys part way through the study and therefore are not marked as 'complete' in the patient flow section, the data they did provide was still used for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I Standard of Care | Arm II Standard of Care Plus Gabapentin
Number analyzed (Participants) | 32 | 39
Participants | 0 | 0
Statistical Analysis 1: Comparison: Arm I Standard of Care vs Arm II Standard of Care Plus Gabapentin; Test type: Superiority; p = 1, Fisher Exact; Odds Ratio (OR) = 1

3. Secondary Outcome: Frequency and Severity of General Systemic Symptoms (Surveys Such as the Neurotoxicity Scale, Profile of Mood States, and Quality of Life Form)
Description: Pain severity will be correlated with frequency and severity of general systemic symptoms. Graphical and descriptive statistical summaries will be generated. Mixed-level general linear modeling will be used. All tests of statistical significance will maintain maximum Type I error of 0.05 (p < 0.05). Baseline pain scores will be included as a covariate in the analyses of the outcome. The General Symptom Survey is a ten item patient reported outcome measure and outcomes were averaged as there is only one item per symptom category. 0 represented no presence of the symptom with a score of 10 representing the most severe symptom.
Time Frame: Up to 3 months post-treatment
Population: Although some patients stopped filling out surveys part way through the study and therefore are not marked as 'complete' in the patient flow section, the data they did provide was still used for analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm I Standard of Care | Arm II Standard of Care Plus Gabapentin
Number analyzed (Participants) | 32 | 39
score on a scale | 1.91 [0.73 to 3.56] | 1.23 [0.45 to 2.79]
Statistical Analysis 1: Comparison: Arm I Standard of Care vs Arm II Standard of Care Plus Gabapentin; Test type: Superiority; p < 0.001, Proportional Odds Regression; Odds Ratio (OR) = 0.371, 95% CI 2-sided [0.244 to 0.597]

ADVERSE EVENTS:
Time Frame: Approximately 3 months after completion of treatment
Arm/Group | Arm I Standard of Care | Arm II Standard of Care Plus Gabapentin
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/41
Other Adverse Events (participants affected / at risk) | 0/38 | 2/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I Standard of Care (N=38) | Arm II Standard of Care Plus Gabapentin (N=41)
Fatigue (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT02480114/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT02480114/Prot_SAP_001.pdf